CLINICAL TRIAL: NCT07030842
Title: Multimodal Deep Learning Models for Predicting Recurrence Pattern in Hepatocellular Carcinoma: A Multicenter Retrospective Development and Validation Study
Brief Title: Precision Recurrence Risk Assessment in Early-stage Hepatocellular Carcinoma
Status: Completed | Type: Observational
Sponsor: Tongji Hospital (Other)
Collaborators: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Wan-Guang Zhang, Professor, Tongji Hospital
Other Study IDs: TJ-IRB20230863
Record Dates: First submitted 2025-06-12; First posted 2025-06-22 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: artificial intelligence; recurrence pattern; multimodal; deep learning
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Hepatectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TJ Cohort (Training/Validation): Internal cohort from Tongji Hospital (2018-2021) used for model training and validation. Includes 462 patients with early-stage HCC who underwent curative resection. Data: preoperative MRI, clinical variables, and postoperative pathology slides. No interventions beyond standard care.
  Interventions: Procedure: liver resection
- SYSMH Cohort (External Test): Independent external test cohort from Sun Yat-sen Memorial Hospital (2021-2022). Includes 117 patients with early-stage HCC meeting identical inclusion criteria. Used to validate generalizability of multimodal DL models. Data anonymized; no additional interventions.
  Interventions: Procedure: liver resection

INTERVENTIONS:
Procedure: liver resection — This is a retrospective observational study analyzing existing clinical data; no experimental interventions were administered. The study evaluates the predictive performance of two deep learning models (preoperative and postoperative) using standard-of-care medical data collected during routine clinical practice, including:
  Preoperative contrast-enhanced MRI scans Postoperative hematoxylin and eosin (H&E)-stained whole slide images Clinical variables (laboratory results, pathology reports, and demographic data)
  All data were collected as part of standard diagnostic and treatment protocols for hepatocellular carcinoma (HCC) patients undergoing liver resection. No additional interventions or modifications to clinical care were implemented for study purposes. The artificial intelligence models were applied to previously acquired, de-identified data to predict aggressive recurrence patterns

SUMMARY:
This retrospective observational study aims to evaluate whether artificial intelligence (AI) models can predict aggressive recurrence in patients who underwent liver resection for early-stage hepatocellular carcinoma (HCC). The main question it seeks to answer is:

Can deep learning models combining preoperative MRI, postoperative pathology slides, and clinical data accurately identify HCC patients at high risk of aggressive recurrence after surgery?

To answer this, the investigators will analyze existing medical data (preoperative MRIs, postoperative whole-slide images, and clinical records) from 579 patients across two medical centers. All data will be anonymized before analysis, and no additional interventions are required from participants.

This study may help clinicians stratify high-risk patients who could benefit from closer surveillance or adjuvant therapies

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent curative liver resection (R0) for pathologically confirmed primary HCC
* BCLC stage 0-A at diagnosis
* Availability of preoperative contrast-enhanced MRI performed within 1 month before surgery
* Availability of postoperative H&E-stained whole slide images (WSIs) with adequate tumor representation
* Complete clinical follow-up data (minimum 2 years if no recurrence)

Exclusion Criteria:

* R1/R2 resection (micro/macroscopically positive margins)
* Missing or poor-quality preoperative MRI (motion artifacts/insufficient contrast enhancement)
* Received neoadjuvant or adjuvant therapy (to avoid treatment confounding)
* Incomplete follow-up (loss to follow-up or missing recurrence status)
* Non-curative procedures (e.g., palliative resection)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This retrospective multicenter study analyzed 579 patients with early-stage hepatocellular carcinoma (HCC) who underwent curative liver resection at two tertiary academic medical centers in China. The study population consisted of:
  Primary Cohort (Training/Validation):
  462 patients from Tongji Hospital (2018-2021)
  External Test Cohort:
  117 patients from Sun Yat-sen Memorial Hospital (2021-2022) All patients met strict inclusion criteria: curative (R0) resection, preoperative MRI within 1 month before surgery, available postoperative pathology slides, and complete follow-up. The population represents typical early-stage HCC patients eligible for surgical resection in endemic areas.
Sampling Method: Non-Probability Sample
Enrollment: 579 (Actual)
Dates: Start 2023-08-25 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Aggressive Recurrence Pattern | 2 years after surgery
  Defined as first recurrence exceeding Milan criteria within 2 years after liver resection.

SECONDARY OUTCOMES:
Recurrence-Free Survival (RFS) | From surgery until first recurrence or July 30, 2024
  Time from surgery date to radiologically confirmed recurrence or last follow-up (until July 30, 2024).
Overall Survival (OS) | From surgery until death or July 30, 2024
  Time from surgery date to death from any cause or last follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China